CLINICAL TRIAL: NCT00460486
Title: Open-Label Phase 3b Clinical Study to Evaluate the Immunogenicity and Safety of FSME-IMMUN 0.5 ml With the First and Second Vaccination Being Administered According to a Rapid Immunization Schedule in Healthy Adults Aged 16 Years or Older
Brief Title: Immunogenicity and Safety Study of FSME-IMMUN 0.5 mL in Adult Subjects Previously Vaccinated According to a Rapid Immunization Schedule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 690601
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Encephalitis, Tick-Borne
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Formaldehyde inactivated, sucrose gradient purified TBE virus antigen, strain Neudörfl

SUMMARY:
The objective of this study is to investigate the immunogenicity and safety of FSME-IMMUN 0.5 ml in two age strata (stratum A: 16 to 49 years, stratum B: > 50 years), with the first and second vaccinations being administered according to a rapid immunization schedule (12 ± 2 days apart). The third vaccination will be administered approximately 6 months after the first dose.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects will be eligible for participation in this study if they:

* Understand the nature of the study, agree to its provisions and provide written informed consent (assent if the subjects is under 18 years of age);
* Provide the written informed consent of their parents / legal guardian (if the subject is under 18 years of age);
* Are aged >= 16 years (from the 16th birthday) at screening;
* Are clinically healthy, (i.e. the physician would have no reservations vaccinating with FSME-IMMUN 0.5 ml outside the scope of a clinical trial);
* Have a negative pregnancy test result at the first medical examination (if female and capable of bearing children);
* Agree to employ adequate birth control measures for the duration of the study (if female and capable of bearing children);
* Agree to keep a Subject Diary.

Exclusion Criteria:

Subjects will be excluded from participation in this study if they:

* Have a history of any previous tick-borne encephalitis (TBE) vaccination;
* Have a history of TBE infection;
* Have a history of infection with or vaccination against other flaviviruses (e.g. dengue fever, yellow fever, Japanese B-encephalitis);
* Have a history of allergic reactions, in particular to one of the components of the vaccine;
* Suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids) that can be expected to influence immunological functions;
* Have a known or suspected problem with drug or alcohol abuse (> 4 liters wine / week or equivalent level of other alcoholic beverages);
* Have donated blood or plasma within 30 days of study entry;
* Have received a blood transfusion or immunoglobulins within 30 days of study entry;
* Are known to be HIV positive (an HIV test is not required specifically for the purpose of this study);
* Are simultaneously participating in another clinical trial including administration of an investigational product;
* Have participated in any other clinical study within six weeks prior to study entry;
* Are pregnant or breastfeeding (if female);
* Are a member of the team conducting this study or are in a dependent relationship with the study investigator. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the investigator.
* Have received any other vaccination within two weeks prior to study entry.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 330
Dates: Start 2006-09; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: Seropositivity rate as determined by Enzyme-Linked Immunosorbent Assay (ELISA) and Neutralization test (NT) at Days 7, 14 and 21 after the second vaccination, in stratum A and B separately, and in the two age strata combined.

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, MD, Principal Investigator — Baxter BioScience
Locations (4):
- Poland (4):
  - Centrum Badan Farmakologii Klinicznej monipol, Krakow
  - Niepubliczny ZOZ "Atarax" s.c., Olsztyn
  - Niepubliczny ZOZ "VITA", Olsztyn
  - "PANTAMED" Sp. z o.o., Olsztyn